CLINICAL TRIAL: NCT06231355
Title: Efficacy of Liposomal Bupivacaine Versus Conventional Bupivacaine for Pain Control in Patients Undergoing Laparoscopic Radical Nephrectomy: A Pilot Randomized Trial
Brief Title: Liposomal vs. Conventional Bupivacaine for Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-553
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Local Anesthetics; Analgesia; Regional Block; Paravertebral Block
Keywords: liposomal bupivacaine; paravertebral block; postoperative pain; nephrectomy
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipo-bupivacaine (Experimental): Paravertebral block is performed with liposomal bupivacaine.
  Interventions: Drug: Performing paravertebral nerve block with lipo-bupivacaine
- Bupivacaine (Active Comparator): Paravertebral block is performed with bupivacaine.
  Interventions: Drug: Performing paravertebral nerve block with bupivacaine

INTERVENTIONS:
Drug: Performing paravertebral nerve block with lipo-bupivacaine — Paravertebral block is performed using liposomal bupivacaine.
  Other Names: 艾恒平 (Ai Heng Ping); Bupivacaine liposome injection
  Arms: Lipo-bupivacaine
Drug: Performing paravertebral nerve block with bupivacaine — Paravertebral block is performed using bupivacaine.
  Other Names: Bupivacaine injection
  Arms: Bupivacaine

SUMMARY:
The goal of this pilot study is to test the hypothesis that liposomal bupivacaine extends the duration of paravertebral block in patients undergoing radical nephrectomy, achieving improved analgesia compared to conventional bupivacaine. The main questions it aims to answer are:

* Area under curve of numeric rating scale of pain from 12 to 72 h after surgery.
* Cumulative opioid consumption during the period of 12 to 72 h after surgery.

DETAILED DESCRIPTION:
Random numbers will be generated by an independent biostatistician in a 1:1 ratio, sealed in sequentially numbered opaque envelopes, and stored by a study coordinator. Only anesthesiologists who perform paravertebral block know group allocation but are not involved in other parts of the trial. Patients, other health-care team members, and investigators for data collection and outcome assessment are masked from group assignments.

Paravertebral block will be performed with either liposomal bupivacaine or plain bupivacaine. The efficacy of nerve block will be assessed every 5 minutes after local anesthetic injection. We will evaluate pain severity, opioid consumption, and occurrence of adverse events at the following timepoints, i.e., end of surgery, 30 minutes after surgery, and 2, 6, 12, 24, 36, 48, 60, and 72 hours after surgery. Additionally, occurrence of complications, quality of recovery, and subjective sleep quality will be assessed during hospital stay after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old.
* Scheduled for laparoscopic-assisted unilateral radical nephrectomy.
* Agree to undergo regional nerve blockade and receive patient-controlled intravenous analgesia after surgery.

Exclusion Criteria:

* Renal cancer with venous thrombus of grade II or higher, or cases that may convert to open surgery.
* Body mass index ≥30 kg/m² or ≤15 kg/m².
* Severe renal dysfunction (serum creatinine >442 μmol/L or requiring renal replacement therapy), severe liver dysfunction (Child-Pugh class C), or American Society of Anesthesiologists class ≥IV.
* Contraindications for deep nerve block, including severe spinal deformity or history of spinal surgery, severe coagulation abnormalities (international normalized ratio >1.7, activated partial thromboplastin time >4 seconds above normal, platelet count <80×10⁹/L), trauma or infection at the planned puncture site, or severe lumbar back pain.
* Chronic opioid dependence and long-term use of various analgesics for more than 3 months.
* Preoperative inability to communicate due to severe dementia, language barriers, or end-stage diseases.
* Preoperative concomitant central nervous system and/or peripheral nervous system diseases.
* Planned endotracheal intubation and admission to the intensive care unit after surgery.
* Known allergy to local anesthetics.
* Other conditions that are deemed unsuitable for trial participation by the attending surgeons or investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
A composite index of pain intensity and opioid consumption (PIOC) between 12 and 72 hours after surgery | Between 12 and 72 hours afer surgery
  The composite index of pain intensity and opioid consumption (PIOC) will be calculated using the area under curve (AUC) of pain intensity and cumulative opioid consumption between 12 and 72 hours in the postoperative period.

SECONDARY OUTCOMES:
Time to onset after paravertebral block | From end of nerve block to initiation of surgery.
  Defined as time interval from end of nerve block to appearance of sensory block.
Time to maximal block after paravertebral block | From end of nerve block to initiation of surgery.
  Defined as time interval from end of nerve block to maximal block).
Extent of paravertebral block | From end of nerve block to 72 hours after surgery.
  Defined as maximal extent of block.
Paravertebral block-related adverse events. | From end of nerve block to initiation of surgery.
  Defined as any unpredictable, unfavourable medical event that is associated with paravertebral block.
A composite index of pain intensity and opioid consumption (PIOC) within 72 hours after surgery. | Up to 72 hours after surgery
  The composite index of pain intensity and opioid consumption (PIOC) will be calculated using the area under curve (AUC) of pain intensity and cumulative opioid consumption between 0.5 and 72 hours in the postoperative period.
Pain intensity within 72 hours after surgery | Up to 72 hours after surgery
  The pain intensity will be assessed both at rest and with movement with the numeric rating scale (an 11-point scale where 0 = no pain, and 10 = the most severe pain) at 0.5, 2, 6, 12, 24, 36, 48, 60, and 72 hours after surgery.
Cumulative opioid consumption within 72 hours after surgery. | Up to 72 hours after surgery
  Cumulative opioid consumption within 72 hours after surgery.

OTHER OUTCOMES:
Patients' satisfaction with pain management. | Up to 3 days after surgery.
  Patients' satisfaction with pain management will be assessed with the numeric rating scale (an 11-point scale where 0 = the most unsatisfied and 10 = the most satisfied.
Incidence of postoperative complications | Up to 30 days after surgery
  Complications are defined as new-onset medical events that are deemed harmful and required therapeutic intervention.
Quality of recovery | At 24 hours after surgery and discharge
  Quality of recovery will be assessed with the QoR-15 questionnaire; scores range from 0 to 150, with higher score indicating better quality of recovery.
Duration of postoperative hospital stay | Up to 30 days after surgery.
  Duration of postoperative hospital stay
Overall in-hospital cost | Up to 30 days after surgery.
  Overall in-hospital cost
Anxiety and depression scores after surgery | At 30 days after surgery.
  Anxiety and depression scores will be assessed with the hospital anxiety and depression scale (HADS, scores range from 0 to 21 for either anxiety or depression, with higher score indicating more severe anxiety and depression).
Postoperative sleep quality | At 1 to 3 days after surgery.
  Postoperative sleep quality will be assessed with the numeric rating scale, scale range from 0 to 10, with higher score indicating better quality of sleep.
Incidence of pain catastrophizing | At 24 hours after surgery and discharge
  Pain catastrophizing will be assessed with the pain catastrophizing scale, scale range from 0 to 52, with higher score(>38) indicating pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ergun M, Berkers AW, van der Jagt MF, Langenhuijsen JF, van Ozdemir-Brunschot D, van der Vliet JA, D'Ancona FC, Warle MC. Components of pain assessment after laparoscopic donor nephrectomy. Acta Anaesthesiol Scand. 2014 Feb;58(2):219-22. doi: 10.1111/aas.12236. Epub 2013 Dec 6. PMID 24308727
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Mathuram Thiyagarajan U, Bagul A, Nicholson ML. Pain management in laparoscopic donor nephrectomy: a review. Pain Res Treat. 2012;2012:201852. doi: 10.1155/2012/201852. Epub 2012 Oct 23. PMID 23150820
- [Background] Simpson JC, Bao X, Agarwala A. Pain Management in Enhanced Recovery after Surgery (ERAS) Protocols. Clin Colon Rectal Surg. 2019 Mar;32(2):121-128. doi: 10.1055/s-0038-1676477. Epub 2019 Feb 28. PMID 30833861
- [Background] Thavaneswaran P, Rudkin GE, Cooter RD, Moyes DG, Perera CL, Maddern GJ. Brief reports: paravertebral block for anesthesia: a systematic review. Anesth Analg. 2010 Jun 1;110(6):1740-4. doi: 10.1213/ANE.0b013e3181da82c8. Epub 2010 May 6. PMID 20448076
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Safa B, Flynn B, McHardy PG, Kiss A, Haslam L, Henry PD, Kaustov L, Choi S. Comparison of the Analgesic Duration of 0.5% Bupivacaine With 1:200,000 Epinephrine Versus 0.5% Ropivacaine Versus 1% Ropivacaine for Low-Volume Ultrasound-Guided Interscalene Brachial Plexus Block: A Randomized Controlled Trial. Anesth Analg. 2021 Apr 1;132(4):1129-1137. doi: 10.1213/ANE.0000000000005373. PMID 33464760
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Malik O, Kaye AD, Kaye A, Belani K, Urman RD. Emerging roles of liposomal bupivacaine in anesthesia practice. J Anaesthesiol Clin Pharmacol. 2017 Apr-Jun;33(2):151-156. doi: 10.4103/joacp.JOACP_375_15. PMID 28781438
- [Background] Pedoto A, Noel J, Park BJ, Amar D. Liposomal Bupivacaine Versus Bupivacaine Hydrochloride for Intercostal Nerve Blockade in Minimally Invasive Thoracic Surgery. J Cardiothorac Vasc Anesth. 2021 May;35(5):1393-1398. doi: 10.1053/j.jvca.2020.11.067. Epub 2020 Dec 2. PMID 33376072
- [Background] Balkhy HH, Arnsdorf S, Krienbring D, Urban J. Liposome Bupivacaine for Postsurgical Analgesia in Patients Undergoing Robotically Assisted Cardiac Surgery. Innovations (Phila). 2015 Nov-Dec;10(6):416-9. doi: 10.1097/IMI.0000000000000190. PMID 26633002
- [Background] Bergese SD, Ramamoorthy S, Patou G, Bramlett K, Gorfine SR, Candiotti KA. Efficacy profile of liposome bupivacaine, a novel formulation of bupivacaine for postsurgical analgesia. J Pain Res. 2012;5:107-16. doi: 10.2147/JPR.S30861. Epub 2012 May 1. PMID 22570563
- [Background] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739
- [Background] NeMoyer RE, Pantin E, Aisner J, Jongco R, Mellender S, Chiricolo A, Moore DF, Langenfeld J. Paravertebral Nerve Block With Liposomal Bupivacaine for Pain Control Following Video-Assisted Thoracoscopic Surgery and Thoracotomy. J Surg Res. 2020 Feb;246:19-25. doi: 10.1016/j.jss.2019.07.093. Epub 2019 Sep 21. PMID 31550671
- [Background] Ilfeld BM, Eisenach JC, Gabriel RA. Clinical Effectiveness of Liposomal Bupivacaine Administered by Infiltration or Peripheral Nerve Block to Treat Postoperative Pain. Anesthesiology. 2021 Feb 1;134(2):283-344. doi: 10.1097/ALN.0000000000003630. PMID 33372949
- [Background] Hussain N, Brull R, Sheehy B, Essandoh MK, Stahl DL, Weaver TE, Abdallah FW. Perineural Liposomal Bupivacaine Is Not Superior to Nonliposomal Bupivacaine for Peripheral Nerve Block Analgesia. Anesthesiology. 2021 Feb 1;134(2):147-164. doi: 10.1097/ALN.0000000000003651. PMID 33372953
- [Background] Dinges HC, Wiesmann T, Otremba B, Wulf H, Eberhart LH, Schubert AK. The analgesic efficacy of liposomal bupivacaine compared with bupivacaine hydrochloride for the prevention of postoperative pain: a systematic review and meta-analysis with trial sequential analysis. Reg Anesth Pain Med. 2021 Jun;46(6):490-498. doi: 10.1136/rapm-2020-102427. Epub 2021 Apr 9. PMID 33837139
- [Background] Kohoutova L, Atlas LY, Buchel C, Buhle JT, Geuter S, Jepma M, Koban L, Krishnan A, Lee DH, Lee S, Roy M, Schafer SM, Schmidt L, Wager TD, Woo CW. Individual variability in brain representations of pain. Nat Neurosci. 2022 Jun;25(6):749-759. doi: 10.1038/s41593-022-01081-x. Epub 2022 May 30. PMID 35637368
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071